CLINICAL TRIAL: NCT00297726
Title: A Prospective Study to Examine the Efficacy of the Arthritis Self Management Program (ASMP) in Patients With Osteoarthritis (OA) in Alberta
Brief Title: A Study to Examine the Efficacy of the Arthritis Self Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Bone and Joint Health Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: PRO-OA-00001
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2006-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis, Ankle; Arthritis; Self-Management
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis | interventions — Self-Management

INTERVENTIONS:
Behavioral: Self-Management Program

SUMMARY:
This study will examine the efficacy of the Arthritis Self Managemnet Program (ASMP)and determine changes in health resource utilization after completeing the ASMP program.

DETAILED DESCRIPTION:
This study will provide an analysis of the efficacy of the Arthritis Self Management Program (ASMP) using both patient administered questionnaires as well as the health utilization data maintained within the administrative databases at Alberta Health and Wellness. This study will also provide other information that has not yet been evaluated in other arthritis self management studies including co-morbidity data and other specific health related utilization information that has not yet been evaluated in other arthritis self management studies including co-morbidity data and other specific health related utilization information as it is recorded in administrative databases, will include a control group and will adjust for potential confounding variables such as sex, age, body mass index (BMI) and stage of disease.

ELIGIBILITY:
Inclusion Criteria:

* OA of the hip and/or knee
* Patient is 18 years of age and over

Exclusion Criteria:

* a concurrent systemic inflammatory disease
* Patient has previously participated in an arthritis self management educational program
* Patient is awaiting total hip or total knee replacement surgery patient has a medical co-morbidity that would render the patient to participate fully in the study procedures, including terminal conditions such as chronic obstructive pulmonary disease, end stage renal disease, heart failure, malignancy with anticipated life expectancy of equal to or less than 2 years
* Patient has been diagnosed with senile dementia or Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2004-10; Study Completion 2006-04

PRIMARY OUTCOMES:
A difference in the WOMAC score of 20 percentage points

SECONDARY OUTCOMES:
A change in health care provider and medication utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril B Frank, MD, Principal Investigator — University of Calgary